CLINICAL TRIAL: NCT03947866
Title: An Observational Clinical Study to Evaluate the Effectiveness of Fixed-dose Combination of eZEtimibe-rosUvaStatin.
Brief Title: Ezetimibe-Rosuvastatin Evaluation Study
Acronym: ZEUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-ROSEZE-EL-160
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Combinations of Drugs; Dependence
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the efficacy of the stable ezetimibe-rosuvastatin combination in patients with primary hypercholesterolemia in achieving the target plasma LCL-C level.

DETAILED DESCRIPTION:
Additional study objectives:

1. Evaluation of the efficacy of the stable ezetimibe-rosuvastatin combination in patients with primary hypercholesterolemia with respect to changes in the rest of the lipid profile (HDL-C, TC, TG).
2. Evaluation of the efficacy of the stable ezetimibe-rosuvastatin combination in patients with primary hypercholesterolemia in altering non-HDL cholesterol (non-HDL - cholesterol) levels.
3. The assessment of the achievement of the LCL-C target of patients receiving the stable ezetimibe-rosuvastatin combination according to their cardiovascular risk category.
4. Assessing patient safety throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have voluntarily consented to participate in the study.
* Adult patients who are already on treatment with the stable combination of ezetimibe-rosuvastatin (Lipopen), at the discretion of the treating physician.
* Adult patient adequately controlled with rosuvastatin and ezetimibe according to ESC / EAS 2019 guidelines.

Exclusion Criteria:

* Patients who have not fully understood the study procedures and have not signed the consent form.
* Patients who are contraindicated for taking the drug according to the Summary of Product Characteristics (MSF) of the study drug.

Hypersensitivity to the active substances or to any of the excipients of Lipopen.

* Pregnancy and breastfeeding.
* Active liver disease involving unexplained, persistent increases in serum transaminases and any increase in serum transaminases that exceeds 3 times the normal upper limit (ULN) or unexplained persistent increases in serum transaminases.
* Patient with severe renal impairment (creatinine clearance <30 ml / min).
* Patient with myopathy
* Patient receiving concomitant treatment with cyclosporine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hyperlcholesterolaemia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
LDL-C | 12 months
  Levels of LDL-C

SECONDARY OUTCOMES:
Lipidemic profile | 12 months
  HDL-C↑ T-CHOL, Triglycerides measurements
Cardiovascular risk factor | 12 months
  Response of patients vs target of total cardiovascular risk to which they belong.
Adverse Events | 12 months
  Number of Adverse Events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Athens University Hospital HIPPOKRATEION, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided